CLINICAL TRIAL: NCT05110794
Title: A Phase 1 Multiple Dose Study to Investigate the Pharmacokinetics, Safety, and Tolerability of LY3502970 in Fed and Fasted Healthy Participants
Brief Title: A Multiple-Dose Study of LY3502970 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18277; J2A-MC-GZGJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06-15

CONDITIONS: Healthy
Keywords: Food; Food Effect
MeSH Terms: interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3502970 (Fed) (Experimental): LY3502970 administered orally to participants who are in a fed state.
  Interventions: Drug: LY3502970
- LY3502970 (Fasted) (Experimental): LY3502970 administered orally to participants who are in a fasted state.
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered Orally.

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LY3502970 is in the bloodstream and how the body handles and eliminates LY3502970 in healthy participants in fed and fasted states. The study will also evaluate the safety and tolerability of LY3502970 in these participants. The study will last up to 49 days excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation.
* Participants with body weight of 45 kilograms (kg) or more and body mass index (BMI) of 18.5 to 35.0 kilograms per meter squared (kg/m²).

Exclusion Criteria:

* Participants who have an abnormal blood pressure and/or pulse rate, deemed to be clinically significant by the investigator at screening.
* Participants who used or intend to use over-the-counter (OTC) or prescription medication and/or herbal/vitamin/traditional medicines or mineral supplements that may affect the safety or objectives of the study, within 14 days prior to dosing and for the duration of the study. Paracetamol and Covid-19 vaccinations are permitted.
* Participants who are currently enrolled in a clinical study involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participants who show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies. A negative test within 6 months of screening would not need to be repeated.
* Participants who show evidence of hepatitis C and/or positive hepatitis C antibody. A negative test within 6 months of screening would not need to be repeated.
* Participants who show evidence of hepatitis B, positive hepatitis B surface antigen, and/or positive hepatitis B core antibody. A negative test within 6 months of screening would not need to be repeated.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3502970 | Predose up to 41 days postdose
  PK: Cmax of LY3502970
PK: Area Under the Concentration-time curve from 0 to 24 hour (AUC0-24) of LY3502970 | Predose up to 41 days postdose
  PK: AUC0-24 of LY3502970
PK: Time to Maximum Observed Concentration (Tmax) of LY3502970 | Predose up to 41 days postdose
  PK: Tmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma X, Liu R, Pratt EJ, Benson CT, Bhattachar SN, Sloop KW. Effect of Food Consumption on the Pharmacokinetics, Safety, and Tolerability of Once-Daily Orally Administered Orforglipron (LY3502970), a Non-peptide GLP-1 Receptor Agonist. Diabetes Ther. 2024 Apr;15(4):819-832. doi: 10.1007/s13300-024-01554-1. Epub 2024 Feb 24. PMID 38402332